CLINICAL TRIAL: NCT00166608
Title: Measurement of Nitrotyrosine Adducts and Cytokines in Acetaminophen Overdose Patients
Brief Title: Cytokines Polymorphisms and Acetaminophen Toxicity
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Laura James, M.D., Arkansas Children's Hospital Research Institute
Other Study IDs: PPRU-10369s; NCT00147407 (obsolete NCT alias)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Drug Toxicity
Keywords: acetaminophen toxicity; liver damage; tylenol overdose
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood sampling

SUMMARY:
Genotyping assays for polymorphisms in the interleukin 10(IL10)gene and the inducible nitric oxide synthase (iNOS) gene will be performed. Genotypes will be compared to the severity of toxicity following overdose.

DETAILED DESCRIPTION:
It was recently reported that IL-10 is protective in Acetaminophen (APAP) toxicity and it down-regulates iNOS production. In an ongoing Pediatric Pharmacology Research Unit (PPRU) Network study, plasma IL-10 levels were higher in patients that developed significant toxicity, as compared to those with minimal hepatic transaminase elevations. In these patients IL-10 elevation is likely a compensatory response to hepatic injury. To further examine the relationship of IL-10 and iNOS in the APAP overdose patients, we will examine genetic variability in the promotor regions of iNOS and IL-10 in patients with APAP overdose. Data from the literature indicate the polymorphisms in the promotor regions of iNOS and IL-10 influence the severity and expression of various diseases. In addition to genotyping for iNOS and IL10 promotor region polymorphisms, plasma levels of nitrotyrosine and IL-10 will be measured in overdose patients.

Blood samples will be obtained from study patients for the analysis of inflammatory cytokines and nitrotyrosine. Blood samples will be obtained at the time of blood sampling for the routine clinical management of the APAP overdose patient. Patients who are hospitalized will have study blood samples drawn at the time daily blood samples are obtained. The sampling will continue daily until the patient is discharged. In addition to blood sampling the following data will be collected: age, gender, race, circumstances of the ingestion, dose of the ingestion, treatment for the ingestion, concomitant therapy, medical history and cigarette use.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any age admitted to a participating site for acetaminophen overdose (acute or chronic).

Exclusion Criteria:

* Patients who are unable to tolerate study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Publication Attached
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2002-12; Primary Completion 2007-05 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To investigate the relationships of cytokines and toxicity in acetaminophen overdose, blood sampleswere collected from patients following acute ingestions of acetaminophen.

CONTACTS AND LOCATIONS:
Overall Officials: Laura James, M.D., Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (7):
- United States (7):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of North Carolina--Chapel Hill, Chapel Hill, North Carolina
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Background] James LP, Simpson PM, Farrar HC, Kearns GL, Wasserman GS, Blumer JL, Reed MD, Sullivan JE, Hinson JA. Cytokines and toxicity in acetaminophen overdose. J Clin Pharmacol. 2005 Oct;45(10):1165-71. doi: 10.1177/0091270005280296. PMID 16172181